CLINICAL TRIAL: NCT05348759
Title: Follow-up Study of the Pulmonary Function and CT Scan Finding in Chronic Kidney Disease Patients After COVID-19 Infection
Brief Title: Pulmonary Function and CT Scan Finding in CKD Patients After COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Other Study IDs: 302/64E
Record Dates: First submitted 2022-04-26; First posted 2022-04-27 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Lung Function Decreased; Xray Complication
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Pulmonary function test — Spirometry was performed by trained nurse at division of pulmonology, Vajira hospital. The forced vital capacity (FVC), forced expiratory volume in first second of exhalation (FEV1), forced mid-expiratory flow (FEF25-75%), and the FEV1/FVC ratio before and after bronchodilators (2 puffs of salbutamol via spacer) were collected in all cases. Total lung capacity (TLC) using the spirometry (Masterscreen PFT, Jaeger, Germany) and diffusion capacity of carbon monoxide was performed in selected case with abnormalities of lung parenchyma found from computed tomography of the chest.
Diagnostic Test: Chest computer scan — High-resolution computed tomography (HRCT) was performed in a single breath-hold on a 128 slice multidetector computed tomography (MDCT) scanner (Philips Healthcare Nederland B.V, Ingenuity 128, Netherlands). HRCT was performed with the patient in the supine position during end-inspiration, supine position during end-expiration, and prone position during end-inspiration with 1 millimeter (mm) slice thickness.

SUMMARY:
COVID-19 is associated with increased morbidity and mortality in patients with chronic kidney disease (CKD) on dialysis. CKD requires particular emphasis during the pandemic due to concern for increased susceptibility to infection from greater use of health facilities in people undergoing maintenance hemodialysis. COVID-19 due to SARS-CoV-2 involves multiple organs and lung injury is one of the most clinical manifestations. The binding of SARS-CoV-2 to the ACE2 receptors at target cells ,including type II pneumocytes ,and alveolar macrophages in the lung could arise into acute systemic inflammatory responses and cytokine storm.The consequentially leading to lung-resident dentritic cells (rDCs) activation, T lymphocytes production and release antiviral cytokines into the alveolar septa and interstitial compartments resulting in diffuse alveolar epithelium destruction,hyaline membrane formation, alveolar septal fibrous proliferation and pulmonary fibrosis.Although it has been reported that subgroups of COVID-19 survivors developed persistent lung parenchymal injury that persisted at least after 6 months 5-6 ,the data in CKD patients has not been reported yet.In addition, a study of pulmonary function test after COVID-19 is needed to be investigated.Thus,we plan to assess pulmonary sequalae of COVID-19 in hemodialysis (HD) patients and pulmonary function test after recovered of infection at least 3 months.

DETAILED DESCRIPTION:
This is the prospective,observational cohort study including CKD stage 5 on hemodialysis who survived acute COVID-19 and presented for clinical follow-up after either mild/moderate or severe COVID-19.The study was conducted at Faculty of Medicine ,Vajira Hospital ,Navamindradhiraj University from June 2022 -September 2022.We adhered to the Declaration of Helsinki,and all patients provided written informed consent before inclusion.Ethics approval was obtained from Institutional Review Board (IRB) prior to start of the study (COA No 302/64 E).

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 5 requiring HD or continuous peritoneal dialysis (CAPD ) for more than 3 months
* Age 18-80 years
* Diagnosis of COVID-19 confirmed by real time polymerase chain reaction (RT-PCR) and recovered for more than3 months previously

Exclusion Criteria:

* patients with history of chronic lung diseases i.e chronic obstructive pulmonary disease (COPD) and restrictive lung disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 end stage renal disease patients requirung renal replacement therapy with history of COVID-19 admitted to Faculty of Medicine, Vajira hospital,Navamindradhiraj University
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Chest CT in ESRD patients after recovered from COVID-19 | 3 months
  Chest CT scan
Pulmonary s function tests in ESRD patients after recovered from COVID-19 | 3 months
  Pulmonary function test

SECONDARY OUTCOMES:
Factors affecting the pumonary sequalae after COVID-19 in CKD patients | 3 months
  oxygen requirement
Factors affecting the pumonary sequalae after COVID-19 in CKD patients | 3 months
  Ventilator needed
Factors affecting the pumonary sequalae after COVID-19 in CKD patients | 3 months
  Interleukin-6 level
Factors affecting the pumonary sequalae after COVID-19 in CKD patients | 3 months
  C-reactive protein level

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine ,Vajira hospital,Navamindradhiraj University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
The investigators planned to share data upon completion of recruitment

REFERENCES:
- [Background] Gagliardi I, Patella G, Michael A, Serra R, Provenzano M, Andreucci M. COVID-19 and the Kidney: From Epidemiology to Clinical Practice. J Clin Med. 2020 Aug 4;9(8):2506. doi: 10.3390/jcm9082506. PMID 32759645
- [Background] Chu H, Chan JF, Wang Y, Yuen TT, Chai Y, Hou Y, Shuai H, Yang D, Hu B, Huang X, Zhang X, Cai JP, Zhou J, Yuan S, Kok KH, To KK, Chan IH, Zhang AJ, Sit KY, Au WK, Yuen KY. Comparative Replication and Immune Activation Profiles of SARS-CoV-2 and SARS-CoV in Human Lungs: An Ex Vivo Study With Implications for the Pathogenesis of COVID-19. Clin Infect Dis. 2020 Sep 12;71(6):1400-1409. doi: 10.1093/cid/ciaa410. PMID 32270184
- [Background] Ooi GC, Khong PL, Muller NL, Yiu WC, Zhou LJ, Ho JC, Lam B, Nicolaou S, Tsang KW. Severe acute respiratory syndrome: temporal lung changes at thin-section CT in 30 patients. Radiology. 2004 Mar;230(3):836-44. doi: 10.1148/radiol.2303030853. PMID 14990845
- [Background] Tharaux PL, Chatziantoniou C, Fakhouri F, Dussaule JC. Angiotensin II activates collagen I gene through a mechanism involving the MAP/ER kinase pathway. Hypertension. 2000 Sep;36(3):330-6. doi: 10.1161/01.hyp.36.3.330. PMID 10988260
- [Background] Hui DS, Wong KT, Ko FW, Tam LS, Chan DP, Woo J, Sung JJ. The 1-year impact of severe acute respiratory syndrome on pulmonary function, exercise capacity, and quality of life in a cohort of survivors. Chest. 2005 Oct;128(4):2247-61. doi: 10.1378/chest.128.4.2247. PMID 16236881
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Derived] Jaturapisanukul S, Yuangtrakul N, Wangcharoenrung D, Kanchanarat K, Radeesri K, Maneerit J, Manomaipiboon A, Rojtangkom K, Ananthanalapa C, Rungrojthanakit S, Thinpangnga P, Alvior J, Trakarnvanich T. Follow-up evaluation of pulmonary function and computed tomography findings in chronic kidney disease patients after COVID-19 infection. PLoS One. 2023 Aug 15;18(8):e0286832. doi: 10.1371/journal.pone.0286832. eCollection 2023. PMID 37582084